CLINICAL TRIAL: NCT01338012
Title: An Open-Label Multicenter Study of Sipuleucel-T in Metastatic Castrate Resistant Prostate Cancer Patients Previously Treated With Sipuleucel-T on Dendreon Study P-11 (NCT00779402)
Brief Title: Sipuleucel-T in Metastatic Castrate Resistant Prostate Cancer
Acronym: mCRPC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative reasons.
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P10-1
Record Dates: First submitted 2011-03-02; First posted 2011-04-19 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: metastatic castrate resistant prostate cancer; prostate cancer; prostate; immune therapy; immunotherapy; vaccine; dendritic cells; antigen-presenting cells; antigen presenting cells; cancer vaccine; prostatic adenocarcinoma; Sipuleucel-T; castration resistant prostate cancer (CRPC); booster; retreatment; immune memory; immune response
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sipuleucel-T (Experimental): Men with metastatic castrate resistant prostate cancer previously treated with sipuleucel-T in the androgen dependent setting in the Dendreon P-11 study. Subjects received one infusion of sipuleucel-T every two weeks for for a total of three infusions.
  Interventions: Biological: sipuleucel-T

INTERVENTIONS:
Biological: sipuleucel-T — Sipuleucel-T is an autologous cellular product consisting of antigen presenting cells (APCs) activated with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF).
  Other Names: PROVENGE, APC8015

SUMMARY:
Multicenter open label, uncontrolled study that enrolled men with metastatic castrate resistant prostate cancer previously treated with sipuleucel-T in the androgen dependent setting in the Dendreon P-11 study. The study was divided into Active and Long Term Follow-up (LTFU) Phases.

DETAILED DESCRIPTION:
Multicenter open label, uncontrolled study that enrolled men with metastatic castrate resistant prostate cancer previously treated with sipuleucel-T in the androgen dependent setting in the Dendreon P-11 study. The study was divided into Active and Long Term Follow-up (LTFU) Phases.

During the Active Phase eligible subjects received one infusion of sipuleucel-T every two weeks for for a total of three infusions. Subjects returned to the clinic for Week 6, Week 10, Month 6, and Month 12 visits. After the Month 12 visit, subjects were to enter the Long Term Follow-up Phase, in which they were contacted every 6 months via telephone.

Study Objectives:

Primary: Evaluate the immune response generated by sipuleucel-T.

Secondary: Evaluate the safety of sipuleucel-T and explore the correlation between sipuleucel-T immune response and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Previously randomized in Dendreon's P-11 study (NCT00779402) and received at least one infusion of sipuleucel-T
* Radiologic evidence of metastasis
* Castrate resistant prostate cancer. Subjects must have current or historical evidence of disease progression concomitant with surgical or medical castration, as demonstrated by PSA progression OR progression of measurable disease OR progression of non-measurable disease
* Castrate level of testosterone (< 50 ng/dL) achieved via medical or surgical castration
* Adequate hematologic function

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Treatment with chemotherapy within 3 months prior to registration
* Treatment with systemic corticosteroids, abiraterone acetate, external beam radiation therapy, or any investigational product for prostate cancer within 28 days prior to registration
* Treatment with commercial sipuleucel-T (Provenge®)
* Current or imminent pathologic long-bone fracture or spinal cord compression
* Known malignancies other than prostate cancer likely to require treatment within 6 months following registration
* A requirement for systemic immunosuppressive therapy for any reason
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to sipuleucel-T or GM-CSF
* Any infection requiring antibiotic therapy or causing fever within 1 week prior to registration
* Any surgery requiring general anesthetic within 28 days prior to registration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Israel, MD, Study Director — Valeant Pharmaceuticals North America LLC
Locations (4):
- United States (4):
  - Orange County Urology Associates, Laguna Hills, California
  - Oregon Health & Science University, Portland, Oregon
  - Virginia Mason Hospital, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sipuleucel-T
Started | 8
Completed | 0
Not Completed | 8
Not completed — Death | 4
Not completed — Study terminated | 4

BASELINE CHARACTERISTICS:
Population: Men who previously participated in Dendreon's P-11 clinical study, received Sipuleucel-T as part of P-11, and who developed metastatic castrate resistant prostate cancer (mCRPC), Safety population includes all subjects who received at least one infusion in the current study (P10-1).
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 74.4 [66 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — ECOG Performance Status is a method used to assess the functional status of a patient. The scale ranges from 0-5. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work; 2=Ambulatory, capable of all self-care but unable to carry out work activities. Up and about >50% of waking hour; 3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead
  Participants
    ECOG 0=Fully Active; No restrictions | 6
    ECOG 1= Restricted Strenuous Activity | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants Enrolled and Treated Prior to Study Termination
Description: Number of study participants that were enrolled and treated in this trial following completion of study P-11 and prior to study termination.
Time Frame: Study duration: date of first subject registration Dec 2011 and date of last subject visit April 2015
Population: This study was terminated early due to administrative reasons. Only eight subjects out of the ninety subjects planned were enrolled and treated. Given the small number of patients enrolled, results should be interpreted with caution.
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: Active phase (screening to Month 12) Follow-up phase: After Month 12 visit to end of study participation
Arm/Group | Sipuleucel-T
All-Cause Mortality (participants affected / at risk) | 4/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T (N=8)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (2)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Device alarm issue (General disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (3)
Peptic ulcer (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sipuleucel-T (N=8)
Eye pain (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Chills (General disorders) | 5 (6)
Fatigue (General disorders) | 4 (9)
Pyrexia (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 1 (3)
Sinusitis (Infections and infestations) | 2 (2)
Citrate toxicity (Injury, poisoning and procedural complications) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Paraesthesia (Nervous system disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to administrative reasons. Only 8 subjects were enrolled and treated. Given the small number of patients enrolled, analyses do not provide reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study will be published and/or presented in an integrated manner reflecting the results observed across all participating center. Accordingly, decisions on timing and content of publications and presentations relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.